CLINICAL TRIAL: NCT04199975
Title: Customized Self-Controlled Power-Driven or Mechanical Orthoses for the Upper Limb - A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Michael Chu Kay MAK, Associate Consultant and Clinical Assistant Professor (Honorary), Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Orthoses_Protocol_v1
Record Dates: First submitted 2019-12-04; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Upper Limb Deformities, Congenital
MeSH Terms: conditions — Upper Extremity Deformities, Congenital | interventions — Orthotic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthoses (Other): Only one single arm in this study
  Interventions: Device: Orthoses

INTERVENTIONS:
Device: Orthoses — Power-Driven or Mechanical Orthoses

SUMMARY:
Patients with congenital or acquired upper limb structural abnormalities and peripheral nerve or brachial plexus palsies have significant loss of function. The use of orthoses may improve function particularly in performing specific tasks for which the orthoses are designed, depending on the patients' deficiencies and needs. The performance of orthoses may be enhanced by being light-weight, motor-driven, and ergonomic.

This pilot, prospective study is designed to test the feasibility and effectiveness of the specially designed orthoses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any congenital or acquired upper limb structural abnormalities
* Patients' condition is not suitable for surgical intervention or patients are not keen for surgical treatment

Exclusion Criteria:

* Patients have no available muscle signal input
* Patients fitted with a pacemaker or an implantable cardioverter defibrillator (ICD) or other implantable electrical devices
* Patients with contact dermatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Pain Score | Baseline
  VAS pain score will be measured
Visual Analogue Scale (VAS) Pain Score | 1-week after
  VAS pain score will be measured
Short-Form Survey (SF-36) | Baseline
  Generic health status instrument to assess quality of life
Short-Form Survey (SF-36) | 1-week after
  Generic health status instrument to assess quality of life
Active and passive range of motion (ROM) | Baseline
  ROM will be measured to determine the joint stiffness
Active and passive range of motion (ROM) | 1-week after
  ROM will be measured to determine the joint stiffness
Disability of Arm, Shoulder and Hand (DASH) questionnaire | Baseline
  Specially designed tool to assess upper extremity disability and symptoms
Disability of Arm, Shoulder and Hand (DASH) questionnaire | 1-week after
  Specially designed tool to assess upper extremity disability and symptoms
Patients' Satisfaction Score | Baseline
  To grade the subjects' satisfaction regarding to their conditions (0=totally not satisfied; 10=fully satisfied)
Patients' Satisfaction Score | 1-week after
  To grade the subjects' satisfaction regarding to their conditions (0=totally not satisfied; 10=fully satisfied)
Grip Strength | Baseline
  Will be measured in kg
Grip Strength | 1-week after
  Will be measured in kg

CONTACTS AND LOCATIONS:
Overall Officials: Chu Kay Michael Mak, FRCSEd(Orth), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No